CLINICAL TRIAL: NCT03529604
Title: Isolation, Quantification and Kinetics of Salivary Ap4A, SCCA and TROP2 in Patients With Oral Cancer and Potentially Malignant Oral Disorders
Brief Title: Salivary Ap4A, SCCA, TROP2 in Oral Cancer Patients
Acronym: OCSALTM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zagreb (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Darko Macan, Professor, PhD, University of Zagreb
Other Study IDs: HRZZ IP-09-2014-9376
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Oral Cavity Squamous Cell Carcinoma; Saliva Altered; Precancerous Lesions
Keywords: Oral Cancer; Potentially Malignant Oral Disorders; Saliva; Squamous cell carcinoma antigen 1; Squamous cell carcinoma antigen 2; Trophoblast cell surface antigen; Diadenosine tetraphosphate
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oral Cancer group: Patients with pathohistologically diagnosed T1 conventional oral squamous cell carcinoma. The investigators will collect saliva from the mouth floor (saliva sampling), measure SCCA1, SCCA2 and TROP2 using ELISA tests and measure Ap4A levels using HPLC.
  Interventions: Other: Saliva sampling; Diagnostic Test: ELISA; Diagnostic Test: HPLC
- PMOD group: Patients with clinically diagnosed leukoplakia, erythroplakia and oral lichen planus. The investigators will collect saliva from the mouth floor (saliva sampling), measure SCCA1, SCCA2 and TROP2 using ELISA tests and measure Ap4A levels using HPLC.
  Interventions: Other: Saliva sampling; Diagnostic Test: ELISA; Diagnostic Test: HPLC
- Control: Age and sex matched subjects. The investigators will collect saliva from the mouth floor (saliva sampling), measure SCCA1, SCCA2 and TROP2 using ELISA tests and measure Ap4A levels using HPLC.
  Interventions: Other: Saliva sampling; Diagnostic Test: ELISA; Diagnostic Test: HPLC

INTERVENTIONS:
Other: Saliva sampling — Saliva was collected from the mouth floor using a specially designed saliva collecting apparatus.
Diagnostic Test: ELISA — Saliva samples will be analyzed using enzyme-linked immunosorbent assay (ELISA) for the detection of SCCA1, SCCA2 and TROP2.
Diagnostic Test: HPLC — High-performance liquid chromatography (HPLC) will be used to measure Ap4A concentrations in saliva.

SUMMARY:
According to the World Health Organization, oral cancer (OC) is the eighth most common cancer in the world with a five year survival rate of 50%.

Oral cancer tumor cells produce biochemical substances, tumor markers, differed from healthy individuals in expression or quantitative ratio, detectable in tissues and/or body fluids.

Saliva, because of its accessibility, proximity and noninvasive approach, presents an ideal tool for the research of oral cancer tumor markers.

The aim of this study will be to isolate, quantify, analyze the role and describe the kinetics of diadenosine tetraphosphate (Ap4A), Squamous Cell Carcinoma associated Antigen (SCCA), Trophoblast cell surface antigen (TROP2) in patients with OC, potentially malignant disorders (PMOD) and age and sex matched control group with a clear medical history.

There are number of studies published on OC tumor markers isolated mostly in serum, however the satisfactory specificity and sensitivity still hasn't been reached.

Liquid chromatography-ion trap-mass spectrometry, Multiple Reaction Monitoring method (LC-IT-MS, MRM) will be developed to isolate and quantify the above mentioned tumor markers. This method has not yet been used to quantify the above mentioned salivary tumor markers. Ap4A and TROP2 have never been isolated from saliva.

The aim is to develop a tumor-specific test with a satisfactory statistical sensitivity and specificity and dynamically measure the levels of tumor markers, before and immediately after therapy - surgery/radiotherapy/chemotherapy or their combination, and during regular follow-up one and two years after surgery. As another novelty, the investigators aim to determine the markers circadian rhythm.

A OC tumor specific test, with satisfactory sensitivity and specificity, would enable earlier OC diagnosis, possibly before the clinical appearance, raise the survival rate of OC patients, enable early diagnosis of recurrence and/or new primary tumors and ensure better post-treatment life-quality.

DETAILED DESCRIPTION:
In the last few years, treatment of oral cancer (OC) showed improvement due to the combined efforts of surgery, radiotherapy and chemotherapy. Nevertheless the long-term survival rate, only marginally improved with a five year survival rate of 50%.

OC is preceded by a preinvasive stage, which may last for many years. Tumor progression in epithelia has been classified as normal, hyperplastic (non-dysplastic), dysplastic carcinoma in situ and invasive carcinoma. The majority of the initial alterations of precancerous and cancerous oral lesions are often non recognizable, even by histopathological examination. The basic biology of initiation and progression of these tumors is still obscure. Carcinogenesis is a process which includes initiation, promotion and progression, driven by accumulation of specific altered genes. Tumor cells produce biochemical substances called tumor markers. Some of these substances found in healthy individuals, but with altered quantitative ratio. Besides the salivary DNA and RNA, other markers are detectable in saliva, such as cell cycle markers (p53, p16 etc.), growth factors (EGF, TGF, etc.), cell surface markers, oxidants and antioxidants and other. Because of its accessibility, non-invasive approach and location proximity, saliva presents an ideal tool for the research of OC tumor markers.

This study will analyze the role of Diadenosine tetraphosphate (Ap4A), Squamous Cell Carcinoma associated Antigen 1 and 2 (SCCA1 and 2) and Trophoblast Cell Surface Antigen (TROP2) in the development of OC.

Ap4A is the only diadenosine polyphosphate that can induce a considerable increase in [Ca2+] in endothelial cells, indicating that its vasoactive effects are comparable to the known effects of arginine vasopressin, angiotensin II and adenosine triphosphate (ATP). Ap4A is a ubiquitous diadenosine polyphosphate signal molecule for DNA replication in mammalian cell.

Level of Ap4A was found to be directly related to the proliferative activity of the cells. It is considered that the Ap4A has an important role in the regulation of cellular growth and division. In the absence of the tumor suppressor gene FHIT (Fragile Histidine Triad), located on the chromosome 3p, Ap4a accumulates and leads to DNA synthesis and multiplication of cells. Loss of heterozygosity of the chromosome 3p is believed to be a common event in the early phase of carcinogenesis.

Ap4A could represent a tumor marker for the early stages of carcinogenesis. Possibly it could indicate carcinogenesis earlier than pathohistological diagnostics. Ap4a has never been isolated in saliva or measured in OC and PMOD patients.

In healthy individuals, SCCA, a glycoprotein, is located inside the cell. In individuals with OC it is released from the cell and thereby, is detectable in serum and saliva. Recent reports have shown that SCCA can influence the invasion or metastasis of cancer cells. However, it remains unclear how SCCA acts to mediate these biological functions. SCCA has already been presented as a potential serum marker for pathologic lymph node metastasis, advanced tumor stage, and an increased rate of distant metastasis in patients with OC, however, never has it been isolated in saliva in OC patients. It has never been measured in patients with PMOD.

The human trophoblast cell-surface antigen, TROP2 (also termed GA733-1, M1S1, EGP-1) is encoded by the TACSTD2 gene, which is mapped to the human chromosome 1p32. TROP2 function and role is still not well understood, although it has previously been suggested that it played a role in growth regulation of cancer cells, as well as in fetal lung formation as a calcium signal transducer. Two studies showed that TROP2 over-expression may emerge as a prognostic tool in patients with oral and laryngeal squamous cell carcinoma. TROP2 antigen has never been isolated or measured in saliva in OC and PMOD patients. OC tumor-specific test will probably have to involve two or all of the above described tumor markers. However, salivary Ap4a alone could present a marker for the earliest stages of OC carcinogenesis. Therefore, it could reveal carcinogenesis before the clinical appearance of OC. The investigators believe that saliva proximity to OC could enable even higher specificity. As another novelty, determining the circadian rhythm of the above mentioned markers should provide more information on their kinetics and role in OC carcinogenesis and rule out any potential confounders, such as the influence of a certain nutritive or the influence of some habits e.g. smoking.

ELIGIBILITY:
Inclusion Criteria:

* pathohistologically confirmed conventional T1 oral squamous cell carcinoma
* clinically diagnosed leukoplakia, erythroplakia and oral lichen planus

Exclusion Criteria:

* ate or drank 2 hours before sampling

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All subjects that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Salivary tumor marker levels before surgery | 1.5.2016.-15.9.2018.
  Salivary tumor marker levels before surgery

SECONDARY OUTCOMES:
Salivary tumor marker levels after surgery | 1.5.2018.-1.9.2019.
  Salivary tumor marker levels after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Darko Macan, PhD, DDS, Principal Investigator — University of Zagreb

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: OFFICIAL PROJECT PAGE — https://ocsaltm.wixsite.com/hrzz-ocsaltm